CLINICAL TRIAL: NCT04465838
Title: A Real World Evidence Study in Chinese Psoriasis Patients
Brief Title: Chinese Psoriasis Real World Evidence Research
Status: Recruiting | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Principal Investigator, Xiaoyong Man, Principal Investigator, Head of Dermatology, Second Affiliated Hospital, School of Medicine, Zhejiang University
Other Study IDs: 2020-354
Record Dates: First submitted 2020-06-26; First posted 2020-07-10 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Psoriasis: This is a non-interventional study (NIS). All the patients diagnosed as psoriasis by the dermatologists in the clinic are included in this study no matter what kind of treatment they adopt.
  Interventions: Other: NIS

INTERVENTIONS:
Other: NIS — This is a non-interventional study (NIS).

SUMMARY:
This research is a multicenter,observational study under real world settings in patients diagnosed as psoriasis by dermatologist in the clinic. As patient's choice of medication should be fully respected, all the patients can choose the treatments they prefer, like phototherapy, traditional systemic therapy or biologics. And the study was conducted to compare the effectiveness among different choices of medication in Chinese psoriasis patients.

DETAILED DESCRIPTION:
Psoriasis is a chronic, recurrent inflammatory disease which is caused by heredity, environment and other factors. The typical clinical manifestation are erythematosquamous lesions, and the disease can progress to involve several organs. In view of its complex pathogenesis, there exists various of treatment of psoriasis like traditional systemic drugs and biologics.

This study is an observational, multi-centre study based on real-world evidence. Inclusion criteria is the patients who visit the clinic diagnosed psoriasis by the dermatologist. There existed no exclusion criteria. Information were most collected by a phone application called "Psoriasis New World".

Primary outcome measure is the percentage of patients who achieved a PASI reduction of 100% (PASI 100). And Psoriasis Area and Severity Index includes scores of erythema, infiltration and desquamation, weighted by area of involvement in each regions (head and neck, upper extremities, trunk, lower extremities), with higher PASI scores indicating worse condition. Also, static Physician Global Assessment (sPGA), static Investigator Global Assessment (sIGA), Body surface area (BSA) and Dermatology Life Quality Index (DLQI) are measured to assess the severity of psoriasis and the change of the disease condition. It is important to monitor all the Adverse Events (AEs) over the whole study. In addition, the laboratory examinations of patients such as liver function are also collected.

ELIGIBILITY:
Inclusion Criteria:

* all the patients diagnosed as psoriasis by dermatologist in clinic.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All the patients diagnosed as psoriasis by dermatologist in clinic were under treatment or willing to be treated.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2020-07-08 (Actual); Primary Completion 2030-07-13 (Estimated); Study Completion 2030-07-30 (Estimated)

PRIMARY OUTCOMES:
The percentage of patients who achieved a PASI reduction of 100% (PASI 100) | 6 months
  Psoriasis Area and Severity Index includes scores of erythema, infiltration and desquamation, weighted by area of involvement in each regions (head and neck, upper extremities, trunk, lower extremities), with higher PASI scores indicating worse condition. The percentage of patients who achieved a PASI reduction of 100% (PASI 100) will be measured.

SECONDARY OUTCOMES:
The percentage of patients who achieved a PASI reduction of 100% (PASI 100) | 6 months and 12 months
  PASI100 represents complete clearance.
The percentage of patients who achieved a PASI reduction of 75% (PASI 75) | 6 months and 12 months
  PASI75 response is the percentage of participants who achieved at least a 75% reduction from baseline in PASI score.
The percentage of patients who achieved a PASI reduction of 50% (PASI 50) | 6 months and 12 months
  PASI50 response is the percentage of participants who achieved at least a 50% reduction from baseline in PASI score.
static Physician Global Assessment (sPGA) = 0 | 6 months and 12 months
  static Physician Global Assessment (sPGA) is an assessment of severity of psoriasis on 5-point scale ranging from 0 to 4.
static Investigator Global Assessment (sIGA) = 0 | 6 months and 12 months
  static Investigator Global Assessment (sIGA) is an assessment of severity of psoriasis on 5-point scale ranging from 0 to 4.
Body surface area (BSA) | 6 months and 12 months
  The percentage of BSA represents the area of involvement, which can be estimated by the entire palm of the patient.
Dermatology Life Quality Index (DLQI) =0 | 6 months and 12 months
  The Dermatology Life Quality Index (DLQI) is a questionnaire used to measure the impact of a skin disease.
Adverse Events (AEs) | Up to 12 months
  Number of patients with adverse events
Visual Analog Scale (VAS) | 6 months and 12 months
  Visual Analog Scale (VAS) is used to measure lesion pruritus from 0 to 10. The higher score is, the greater discomfortableness participant has.

CONTACTS AND LOCATIONS:
Locations (29):
- China (29):
  - Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang
  - Beijing Children's Hospital Affiliated to Capital Medical University, Beijing
  - the First Affiliated Hospital of Chongqing Medical University, Chongqing
  - the First Affiliated Hospital of Fujian Medical University, Fujian
  - General Hospital of Lanzhou Military Region, Gansu
  - Sun Yat-sen Memorial Hospital, Guangdong
  - The Peoples' Hospital of Guangxi Zhuang Autonomous Region, Guangxi
  - the Affiliated Hospital of Guizhou Medical University, Guizhou
  - The Fifth People's Hospital of Hainan Province, Hainan
  - the First Hospital of Hebei Medical University, Hebei
  - the Second Affiliated Hospital of Harbin Medical Unviersity, Heilongjiang
  - Henan Provincial Peoples' Hospital, Henan
  - the Affiliated Hospital of Inner Mongolia Medical University, Hohhot
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Hubei
  - Xiangya Hospital, Central South University, Hunan
  - the Second Affiliated Hospital of Nanchang University, Jiangxi
  - Yanbian University Hospital, Jilin
  - Institute of Dermatology, Chinese Academy of Medical Sciences, Nanjing
  - Xining First Hospital, Qinghai
  - Shandong Provincial Hospital for Skin Diseases, Shandong
  - Shanghai Dermatology Hospital, Shanghai
  - Taiyuan Central Hospital, Shanxi
  - the Second Affiliated Hospital of Xi'an Jiaotong University, Shanxi
  - the First hospital of China Medical University, Shenyang
  - Sichuan Provincial People's Hospital, Sichuan
  - Tianjin Academy of Traditional Chinese Medicine Affiliated Hospital, Tianjin
  - First Affiliated Hospital, School of Medicine, Shihezi University, Xinjiang
  - General Hospital of Ningxia Medical University, Yinchuan
  - the Second Affiliated Hospital of Kunming Medical University, Yunnan

IPD SHARING:
Plan to Share IPD: Undecided